CLINICAL TRIAL: NCT07216248
Title: A Phase II Randomized, Decentralized, De-escalation Study in Patients With Metastatic Hormone-Sensitive Prostate Cancer Achieving Optimal PSA Response (OPTIMAS)
Brief Title: Optimal PSA Triggered Individual Management of Androgen Sensitive Prostate Cancer
Acronym: OPTIMAS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI194008
Record Dates: First submitted 2025-09-30; First posted 2025-10-14 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer (mHSPC)
MeSH Terms: interventions — relugolix; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A: Arm 1 (Active Comparator): INDUCTION (Step 1): Participants will receive continuous treatment with relugolix + an androgen receptor pathway inhibitor (ARPI).
  After 6-12 months of continuous treatment, participants whose PSA is ≤ 0.2 ng/mL and who have completed step two registration will be randomized to one of two treatment arms:
  • Cohort A: Arm 1 will continue standard-of-care, continuous treatment with relugolix or androgen deprivation therapy (ADT) + ARPI per clinical investigator.
  Interventions: Drug: relugolix + ARPI; Drug: relugolix or androgen deprivation therapy (ADT) + ARPI
- Cohort A: Arm 2 (Experimental): INDUCTION (Step 1): Participants will receive continuous treatment with relugolix + an androgen receptor pathway inhibitor (ARPI).
  After 6-12 months of continuous treatment, participants whose PSA is ≤ 0.2 ng/mL and who have completed step two registration will be randomized to one of two treatment arms:
  • Cohort A: Arm 2 will receive intermittent treatment with relugolix + ARPI.
  Interventions: Drug: relugolix + ARPI; Drug: relugolix + ARPI.
- Cohort B (Experimental): Participants who have achieved PSA ≤ 0.2 ng/mL are eligible and will receive intermittent treatment with relugolix + ARPI.
  Interventions: Drug: Intermittent- Relugolix or androgen deprivation therapy (ADT) + ARPI

INTERVENTIONS:
Drug: relugolix + ARPI — Step 1: Continuous treatment with relugolix + ARPI
  Arms: Cohort A: Arm 1; Cohort A: Arm 2
Drug: Intermittent- Relugolix or androgen deprivation therapy (ADT) + ARPI — Intermittent treatment with relugolix + ARPI.
  Arms: Cohort B
Drug: relugolix or androgen deprivation therapy (ADT) + ARPI — Step 2: Standard-of-care, continuous treatment with relugolix or androgen deprivation therapy (ADT) + ARPI.
  Arms: Cohort A: Arm 1
Drug: relugolix + ARPI. — Step 2: Intermittent treatment with relugolix + ARPI.
  Arms: Cohort A: Arm 2

SUMMARY:
The purpose of this study is to evaluate intermittent relugolix + androgen receptor pathway inhibitor (ARPI) in patients with metastatic hormone-sensitive prostate cancer (mHSPC) achieving optimal PSA response.

ELIGIBILITY:
Inclusion Criteria:

Cohort A Eligibility (Step 1 Registration)

* Participant aged ≥ 18 years
* Hormone-sensitive prostate cancer with histologically/cytologically confirmed adenocarcinoma without small cell histology.
* Metastasis detected any time prior to study registration on conventional or functional imaging as determined by the treating investigator and can be of any site.
* Baseline testosterone >50 ng/dl before start of therapy for metastatic disease
* PSA ≥ 1 ng/mL
* ECOG Performance Status ≤ 2
* Eligible to receive standard of care treatment with relugolix and APRI per clinical investigator.
* Participants with a sexual partner of childbearing potential must agree to use a highly effective method of contraception requirements as described in Section 5.5.1.

  * If the risk of seminal transfer from the participant is present, the participant must agree to use a condom during sexual intercourse as described in Section 5.5.2.
  * Participants must agree not to donate sperm from the start of study therapy until 3 months after the last dose of study therapy.
* Clinically significant adverse effects from any prior oncologic treatment (e.g. prior surgery, radiotherapy, or other antineoplastic therapy) must have resolved or have been determined to be clinically stable per the Investigator.
* Has access to a smartphone and wireless services and is able to download and navigate study specific applications.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Cohort A Eligibility (Step 2 Registration) -PSA ≤ 0.2 ng/mL after 6-12 months of relugolix and androgen receptor pathway inhibitor treatment. Androgen receptor pathway inhibitor includes abiraterone, enzalutamide, apalutamide, darolutamide or similar drugs.

Cohort B Eligibility

* Participant aged ≥ 18 years
* Hormone-sensitive prostate cancer with histologically/cytologically confirmed adenocarcinoma without small cell histology.
* Metastasis detected any time prior to study registration on conventional or functional imaging as determined by clinical investigator and can be of any site.
* PSA ≤ 0.2 ng/mL after treatment with androgen deprivation therapy or androgen receptor pathway inhibitor treatment or both of any duration. Androgen deprivation therapy in this context includes gonadotropin-releasing hormone agonists and antagonists. Androgen receptor pathway inhibitors include abiraterone, enzalutamide, apalutamide, darolutamide or similar drugs.
* Eligible to receive standard of care treatment with relugolix and APRI per clinical investigator.
* Participants with a sexual partner of childbearing potential must agree to use a highly effective method of contraception requirements as described in Section 5.5.1.

  * If the risk of seminal transfer from the participant is present, the participant must agree to use a condom during sexual intercourse as described in Section 5.5.2.
  * Participants must agree not to donate sperm from the start of study therapy until 3 months after the last dose of study therapy.
* Has access to a smartphone and wireless services and is able to download and navigate study specific applications.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

Cohort A Eligibility (Step 1 Registration)

* Participant received androgen deprivation therapy (defined as leuprolide or surgical castration) for metastatic hormone-sensitive prostate cancer.
* The diagnosis of another malignancy which, in the opinion of the Investigator, is likely to negatively impact the participant's safety or ability to participate in the study.
* Known brain metastases or cranial epidural disease.

  --Note: Brain metastases or cranial epidural disease adequately treated with radiotherapy and/or surgery and stable for at least 4 weeks before the first dose of study treatment will be allowed on trial. Participants must be neurologically stable and receiving a stable or decreasing corticosteroid dose at the time of study entry.
* Current evidence of uncontrolled, significant intercurrent illness, infection, non-compliance or other safety concerns which may affect clinical trial participation.
* Medical, psychiatric, cognitive, or other conditions that may compromise the participant's ability to understand the participant information, give informed consent, comply with the study protocol or complete the study.
* Known prior severe hypersensitivity to investigational product or any component in its formulations (CTCAE v5.0 Grade ≥ 3).
* Participants taking prohibited medications as described in Section 6.6.2.

Cohort A Eligibility (Step 2 Registration)

* Receiving other systemic anti-cancer therapy for prostate cancer. Prior treatment before Step 2 registration is allowed.
* Progression to metastatic castration-resistant prostate cancer per clinical investigator.
* The diagnosis of another malignancy which, in the opinion of the Investigator, is likely to negatively impact the participant's safety or ability to participate in the study.
* Participants taking prohibited medications as described in Section 6.6.2.

Cohort B Eligibility

* Receiving other systemic anti-cancer therapy for prostate cancer.
* History of surgical castration.
* The diagnosis of another malignancy which, in the opinion of the Investigator, is likely to negatively impact the participant's safety or ability to participate in the study.
* Known brain metastases or cranial epidural disease.

  --Note: Brain metastases or cranial epidural disease adequately treated with radiotherapy and/or surgery and stable for at least 4 weeks before the first dose of study treatment will be allowed on trial. Participants must be neurologically stable and receiving a stable or decreasing corticosteroid dose at the time of study entry
* Current evidence of uncontrolled, significant intercurrent illness, infection, compliance or other safety concerns which may affect clinical trial participation.
* Medical, psychiatric, cognitive, or other conditions that may compromise the participant's ability to understand the participant information, give informed consent, comply with the study protocol or complete the study.
* Known prior severe hypersensitivity to investigational product or any component in its formulations (CTCAE v5.0 Grade ≥ 3).
* Participants taking prohibited medications as described in Section 6.6.1.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Cohort A: Brief Fatigue Inventory (BFI) score 6 months after randomization. | 6 months
  To assess the difference in fatigue 6 months after randomization in patients with mHSPC achieving optimal PSA response on intermittent relugolix + ARPI versus continuous relugolix/ADT + ARPI. Scored from 0 (no Fatigue) to 10 (as bad as you can imagine), and 0 (Does not interfere) to 10 (Completely Interferes).
Cohort B: Progression-free survival (PFS) as defined as the time from intermittent study initiation (first treatment break) to the time of documented disease progression or death from any cause at one year. | 12 months
  To assess PFS in patients with mHSPC on intermittent relugolix + ARPI at one year.

SECONDARY OUTCOMES:
Changes in health-related quality of life as measured by the European Organisation for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC-QLQC30). | 13 months
  To evaluate treatment effects on patient-reported outcomes (PROs). EORTC-QLQC30 scored from 1 (not at all)- 4 (very much).
Changes in health-related quality of life as measured by the European Organisation for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC-QLQ-PR25). | 13 months
  To evaluate treatment effects on patient-reported outcomes (PROs). EORTC-QLQ-PR25 scored from 1 (not at all)- 4 (very much).
Sexual function improvement in those with intact sexual function at baseline as measured by the European Organisation for Research and Treatment of Cancer Quality of Life Core Questionnaire. | 13 months
  To evaluate treatment effects on patient-reported outcomes (PROs). EORTC-QLQ-PR25, question 52-55.Scored from 1 (not at all)- 4 (very much).
Changes in severity of hot flashes as measured by the Hot Flash Related Daily Interference Scale (HFRDIS). | 13 months
  To evaluate treatment effects on patient-reported outcomes (PROs). HFRDIS scored 0 (did not interfere to 10 (completely interfered).
Changes in cognitive function as measured by the PROMIS-Cognitive function Short Form 8a. | 13 months
  To evaluate treatment effects on patient-reported outcomes (PROs). PROMIS-Cognitive function Short Form 8a scored 5 (Never)- 1 (very often- Several times a day).
Change from baseline over time in each PRO, including time to recovery and deterioration in the intermittent arm with treatment break and start. | 2 years
  To evaluate treatment effects on patient-reported outcomes (PROs).
Time to metastatic castration-resistant prostate cancer. | 12 months
  Cohort A: To determine if intermittent relugolix + ARPI will provide similar efficacy as continuous relugolix/ADT + ARPI in clinically relevant endpoints in participants with mHSPC who reached PSA ≤0.2 ng/mL after 6-12 months of relugolix+ARPI treatment.
  Cohort B: To evaluate the treatment efficacy of intermittent relugolix + ARPI.
Overall survival and prostate cancer-specific survival at 3 years from the date of randomization. | 12 months
  Cohort A: To determine if intermittent relugolix + ARPI will provide similar efficacy as continuous relugolix/ADT + ARPI in clinically relevant endpoints in participants with mHSPC who reached PSA ≤0.2 ng/mL after 6-12 months of relugolix+ARPI treatment.
  Cohort B: Change from baseline over time in each PRO, including time to recovery and deterioration in intermittent arm with treatment break and start.
Time to systemic treatment change. | 12 months
  To determine if intermittent relugolix + ARPI will provide similar efficacy as continuous relugolix/ADT + ARPI in clinically relevant endpoints in participants with mHSPC who reached PSA ≤0.2 ng/mL after 6-12 months of relugolix+ARPI treatment
Duration of time on treatment | 12 months
  Cohort A: To determine if intermittent relugolix + ARPI will provide similar efficacy as continuous relugolix/ADT + ARPI in clinically relevant endpoints in participants with mHSPC who reached PSA ≤0.2 ng/mL after 6-12 months of relugolix+ARPI treatment.
  Cohort B: To evaluate the treatment efficacy of intermittent relugolix + ARPI.
Time to first treatment restart | 12 months
  Cohort A: To determine if intermittent relugolix + ARPI will provide similar efficacy as continuous relugolix/ADT + ARPI in clinically relevant endpoints in participants with mHSPC who reached PSA ≤0.2 ng/mL after 6-12 months of relugolix+ARPI treatment.
  Cohort B: To evaluate the treatment efficacy of intermittent relugolix + ARPI.
Duration of time with testosterone < 50 ng/mL | 12 months
  Cohort A: To determine if intermittent relugolix + ARPI will provide similar efficacy as continuous relugolix/ADT + ARPI in clinically relevant endpoints in participants with mHSPC who reached PSA ≤0.2 ng/mL after 6-12 months of relugolix+ARPI treatment.
  Cohort B: To evaluate the treatment efficacy of intermittent relugolix + ARPI.
Testosterone-linked outcomes (time to recovery of testosterone ≥50 ng/dL; time to recovery of testosterone to baseline [≥screening testosterone level]). | 12 months
  Cohort A: To determine if intermittent relugolix + ARPI will provide similar efficacy as continuous relugolix/ADT + ARPI in clinically relevant endpoints in participants with mHSPC who reached PSA ≤0.2 ng/mL after 6-12 months of relugolix+ARPI treatment.
  Cohort B: To evaluate the treatment efficacy of intermittent relugolix + ARPI.
Duration of time to recovery of testosterone to normal range [>300 ng/dL]). | 12 months
  Cohort A: To determine if intermittent relugolix + ARPI will provide similar efficacy as continuous relugolix/ADT + ARPI in clinically relevant endpoints in participants with mHSPC who reached PSA ≤0.2 ng/mL after 6-12 months of relugolix+ARPI treatment.
  Cohort B: To evaluate the treatment efficacy of intermittent relugolix + ARPI.
The proportion of participants achieving a treatment-free interval (TFI) of at least one year from the time of registration and median TFI. | 12 months
  To assess the TFI at one year in patients achieving optimal PSA response.
Change in Brief Fatigue Inventory (BFI) score from baseline to 6 months after registration. | 6 months
  To assess the change in quality of life measures from baseline. BFI Scored from 0 (no Fatigue) to 10 (as bad as you can imagine), and 0 (Does not interfere) to 10 (Completely Interferes).
Changes in cognitive function as measured by the PROMIS-Cognitive Function Short Form 8a. | 13 months
  To assess the change in quality of life measures from baseline. PROMIS-Cognitive function Short Form 8a scored 5 (Never)- 1 (very often- Several times a day).
Change from baseline over time in each PRO, including time to recovery and deterioration in intermittent arm with treatment break and start. | 13 months
  To assess the change in quality of life measures from baseline.
Overall survival and prostate cancer specific survival at 3 years from the date of randomization. | 3 years
  To evaluate the treatment efficacy of intermittent relugolix + ARPI.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States